CLINICAL TRIAL: NCT00981786
Title: Quality of 24-hour Intraocular Pressure Control Obtained With the Brinzolamide/Timolol Fixed Combination Compared With the Brimonidine/Timolol Fixed Combination When Added to Travoprost Monotherapy in Subjects With Open-angle Glaucoma
Brief Title: 24-Hour Intraocular Pressure With Brinzolamide/Timolol Versus Brimonidine/Timolol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A434
Record Dates: First submitted 2009-09-16; First posted 2009-09-22 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Glaucoma
Keywords: 24-hour IOP control; brinzolamide/timolol; brimonidine/timolol; travoprost
MeSH Terms: conditions — Glaucoma | interventions — Brimonidine Tartrate; Brimonidine Tartrate, Timolol Maleate Drug Combination; brinzolamide; Azarga

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brinzolamide/Timolol therapy (Active Comparator): Chronic therapy for 3 months with brinzolamide/timolol drops given twice daily added to travoprost drops
  Interventions: Drug: Brimonidine/timolol fixed combination drops added to travoprost; Drug: Brinzolamide/timolol fixed combination drops added to travoprost
- Brimonidine/Timolol therapy (Active Comparator): Chronic therapy for 3 months with brimonidine/timolol drops given twice daily added to travoprost drops
  Interventions: Drug: Brimonidine/timolol fixed combination drops added to travoprost; Drug: Brinzolamide/timolol fixed combination drops added to travoprost

INTERVENTIONS:
Drug: Brimonidine/timolol fixed combination drops added to travoprost — twice daily administration
  Other Names: Combigan
Drug: Brinzolamide/timolol fixed combination drops added to travoprost — twice daily dosing
  Other Names: Azarga

SUMMARY:
The proposed crossover study will compare for the first time the quality of 24-hour intraocular pressure control with the combination of travoprost and brinzolamide/timolol compared with travoprost and brimonidine/timolol in glaucoma patients insufficiently controlled with travoprost. This comparison may determine the real efficacy of the two fixed combinations when added to the prostaglandin. The design of the proposed study should facilitate a better understanding of the role of these medications in glaucoma management.

ELIGIBILITY:
Inclusion Criteria:

* Patient has open-angle glaucoma and is older than 29 years
* Patients should exhibit typical disc, or field changes and an untreated morning IOP greater than 25 mm Hg
* Patients are treated for at least 3 months with travoprost and should have demonstrated at least a 20% morning IOP reduction
* Patient deemed by PI to require adjunctive therapy to obtain desired target IOP
* Patient should exhibit IOP greater than 18 mm Hg on travoprost monotherapy (2 separate IOP readings at 10:00)
* Patient has mild to moderate glaucoma (field loss more than 16 dB; cupping 0.8 or less)
* Distance best corrected Snellen visual acuity at least 0.1
* No contraindications to travoprost, brimonidine, brinzolamide and β-blockers
* No history of lack of response (<10% morning IOP reduction) to any medication
* Patient can understand the instructions and adhere to medications

Exclusion Criteria:

* Female patient of childbearing potential or lactating mother
* History of trauma, inflammation, surgery
* History of past use of steroids (within 2 months), severe dry eyes and use of contact lenses
* Signs of ocular infection, except blepharitis
* Evidence of corneal abnormality that may affect IOP measurements etc
* Closed angle
* History of non-compliance

Ages: 29 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Mean 24-hour intraocular pressure | 3 months

SECONDARY OUTCOMES:
Fluctuation of 24-hour intraocular pressure | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios G Konstas, MD, PhD, Principal Investigator — Glaucoma Unit, 1st University Department of Ophthalmology

IPD SHARING:
Plan to Share IPD: No